CLINICAL TRIAL: NCT01815359
Title: ICARuS (Intraperitoneal Chemotherapy After cytoReductive Surgery): A Multi-center, Randomized Phase II Trial of Early Post-operative Intraperitoneal Chemotherapy (EPIC) and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) After Optimal Cytoreductive Surgery (CRS) for Neoplasms of the Appendix, Colon or Rectum With Isolated Peritoneal Metastasis
Brief Title: ICARuS Post-operative Intraperitoneal Chemotherapy (EPIC) and Hyperthermic Intraperitoneal Chemotherapy (HIPEC) After Optimal Cytoreductive Surgery (CRS) for Neoplasms of the Appendix, Colon or Rectum With Isolated Peritoneal Metastasis
Acronym: ICARuS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The Cleveland Clinic (Other); Brigham and Women's Hospital (Other); University of Miami (Other); University of Pittsburgh Medical Center (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-289
Record Dates: First submitted 2013-03-13; First posted 2013-03-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Appendix Cancer; Colorectal Cancer
Keywords: ICARuS; Intraperitoneal Chemotherapy; hyperthermic intraperitoneal chemotherapy; Optimal Surgical Debulking; Leucovorin; Floxuridine (FUDR); Mitomycin; 12-289
MeSH Terms: conditions — Appendiceal Neoplasms; Colorectal Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy; Mitomycin; Floxuridine; Leucovorin

STUDY DESIGN:
Intervention Model Description: After the initial 212 patients are accrued, the final 70 patients will be accrued to only the appendiceal cohorts

ARMS (4):
- Appendiceal, no chemotherapy within 6 months prior to surgery (Experimental): First, patients will be stratified by previous systemic chemotherapy and by the organ of origin as determined by the PI or Co-PI.
  1. Exposure to chemotherapy in the prior 6 months vs. no such exposure
  2. Appendix vs. Colon or Rectum Then, patients will be randomly assigned in the operating room, by envelope, to either HIPEC (Group A) or EPIC (Group B) after the operating surgeon determines that the patient is optimally cytoreduced to nodules no greater than 2.5mm.
  Interventions: Procedure: Cytoreductive Surgery; Drug: HIPEC with Mitomycin-C; Drug: EPIC with FUDR and Leucovorin
- Appendiceal, chemotherapy within 6 months prior to surgery (Experimental): First, patients will be stratified by previous systemic chemotherapy and by the organ of origin as determined by the PI or Co-PI.
  1. Exposure to chemotherapy in the prior 6 months vs. no such exposure
  2. Appendix vs. Colon or Rectum • Then, patients will be randomly assigned in the operating room, by envelope, to either HIPEC (Group A) or EPIC (Group B) after the operating surgeon determines that the patient is optimally cytoreduced to nodules no greater than 2.5mm.
  Interventions: Procedure: Cytoreductive Surgery; Drug: HIPEC with Mitomycin-C; Drug: EPIC with FUDR and Leucovorin
- Colorectal, no chemotherapy within 6 months prior to surgery (Experimental): First, patients will be stratified by previous systemic chemotherapy and by the organ of origin as determined by the PI or Co-PI.
  1. Exposure to chemotherapy in the prior 6 months vs. no such exposure
  2. Appendix vs. Colon or Rectum • Then, patients will be randomly assigned in the operating room, by envelope, to either HIPEC (Group A) or EPIC (Group B) after the operating surgeon determines that the patient is optimally cytoreduced to nodules no greater than 2.5mm.
  Interventions: Procedure: Cytoreductive Surgery; Drug: HIPEC with Mitomycin-C; Drug: EPIC with FUDR and Leucovorin
- Colorectal, chemotherapy within 6 months prior to surgery (Experimental): First, patients will be stratified by previous systemic chemotherapy and by the organ of origin as determined by the PI or Co-PI.
  1. Exposure to chemotherapy in the prior 6 months vs. no such exposure
  2. Appendix vs. Colon or Rectum • Then, patients will be randomly assigned in the operating room, by envelope, to either HIPEC (Group A) or EPIC (Group B) after the operating surgeon determines that the patient is optimally cytoreduced to nodules no greater than 2.5mm.
  Interventions: Procedure: Cytoreductive Surgery; Drug: HIPEC with Mitomycin-C; Drug: EPIC with FUDR and Leucovorin

INTERVENTIONS:
Procedure: Cytoreductive Surgery — Optimal Surgical Debulking
Drug: HIPEC with Mitomycin-C
Drug: EPIC with FUDR and Leucovorin

SUMMARY:
This is the first randomized trial comparing Early post-operative intraperitoneal chemotherapy (EPIC) and hyperthermic intraperitoneal chemotherapy (HIPEC) for appendiceal and colorectal cancer. The purpose of this study is to find out what effects, good and/or bad, EPIC and HIPEC after cytoreductive surgery have on the patient and the appendiceal, rectal or colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age 18 years or older, both genders.
* Clinical diagnosis of appendiceal or colorectal neoplasm with peritoneal mucinosis or metastasis.
* Patient must be planning to undergo complete cytoreduction of all peritoneal disease.
* ECOG performance status ≤ 1.
* Hematology: ANC ≥ 1,500/ μL; Platelets > 75,000/ μL.
* Adequate Renal function Creatinine <1.5 x the upper limit of normal (ULN) or calculated creatinine clearance of ≥ 50ml/min.
* Adequate Hepatic function: Bilirubin less than 1.5mg/dL; (except in patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0mg/dL).
* Women with childbearing potential who are negative for pregnancy test (urine or blood) and who agree to use effective contraceptive method. Reliable contraception should be used from trial screening and must be continued throughout the study. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant.
* A man participating in this study must agree to utilize reliable barrier form of contraception for the duration of the study.
* Signed and dated written informed consent to participate in this clinical trial must be obtained prior to any study procedure.
* Subjects with a history of endometrial cancer are eligible only if they presented with a stage lower than 1A and if the histology was a subtype other than poorly differentiated.

Exclusion Criteria:

* Subjects who have previously undergone intraperitoneal chemotherapy.
* Subjects with classical carcinoid
* Tumors of low malignant potential
* Other prior malignancies, except for cured non-melanoma skin cancer, curatively treated in situ carcinoma of the cervix, adequately treated malignancies for which there has been no evidence of activity for more than 3 years or indolent tumors for which observation over three years is a reasonable option.
* Presence of clinically apparent or suspected metastasis to sites other than lymph nodes or peritoneal surfaces.
* Women who are pregnant or lactating.
* Subjects with a condition which may interfere with the subjects' ability to understand the requirements of the study.
* Active coronary artery disease (defined as unstable angina or a positive cardiac stress test).
* Subjects with a history of coronary artery disease may be included if they have had a normal stress test within 60 days of enrollment and/or were cleared by MSK cardiology.
* Uncontrolled hypertension defined as >140/90 and not cleared for surgery at the time of consent.
* New York Heart Association (NYHA) Class II or higher Congestive heart failure.
* Restrictive or obstructive pulmonary disease that would limit study compliance or place the patient at unacceptable risk for participation in the study.
* History of cerebrovascular disease. that would limit study compliance or place the patient at unacceptable risk for participation in the study.
* Subjects with other concurrent severe medical problems unrelated to the malignancy that would significantly limit full compliance with the study or places them at an unacceptable risk for participation in the study.
* Patients with known floxuridine, leucovorin ,or mitomycin allergy.
* Evidence of extensive intraperitoneal adhesions at the time of surgery which prohibits intraperitoneal therapy, as determined by the operating surgeon.
* Any condition that would preclude the ability to deliver appropriate IP therapy.
* Use of an oral medication, lacking a suitable non-oral substitute, that if held for up to ten days, would be felt an unacceptable risk by the investigator.
* Life expectancy < 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2013-03; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years
  Documentation of tumor recurrence will be made based on surveillance CT/PET CT scans at time points as determined by attending radiologist, with clinical correlation from the treating physician.

SECONDARY OUTCOMES:
surgical toxicity grade 3 to 5 | up to 60 days
  We will evaluate toxicity up to 30 days postoperatively for any surgical Grade 3-5 complications/toxicites or chemotherapy related Grade 4 or 5 toxicities. Surgical morbidity will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
chemotherapy toxicity grade 3 to 5 | up to 60 days
  We will evaluate toxicity up to 30 days postoperatively for any surgical Grade 3-5 complications/toxicities or chemotherapy related Grade 4 or 5 toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Garrett Nash, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of Miami, Miami, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow up), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow up), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/